CLINICAL TRIAL: NCT04373005
Title: A Research Platform to Screen Patients in Oncology and Assess Impact - RESPONSE
Brief Title: Screening of Cancer Patients to Assess Impact of COVID-19
Status: Terminated | Type: Observational
Why Stopped: Participants were not testing positive for COVID-19 and were not returning onsite for visits.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: U-DEPLOY: RESPONSE; CAPCR 20-5337 (Other: University Health Network)
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Covid-19; Cancer
MeSH Terms: conditions — COVID-19; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nasopharyngeal (NP) swabs: NP swabs:
  * At the time of consent
  * 3-6 weeks after starting cancer treatment (for patients whose treatment has yet not started) or 3-6 weeks after first swab (for patients already on treatment)
  * 3 months after second swab
  * 6 months after second swab
  * 12 months after second swab
  Interventions: Diagnostic Test: Nasopharyngeal (NP) swab

INTERVENTIONS:
Diagnostic Test: Nasopharyngeal (NP) swab — A dry swab will be inserted through one nostril straight towards the back of the nasal passage and rotated gently before the swab is removed.

SUMMARY:
The purpose of this study is to investigate the impact of COVID -19 in the cancer patient population. This will be done by looking at the rate of asymptomatic COVID-19 infection in cancer patients receiving cancer therapy, as well as their immune response.

This is a sub-study of the U-DEPLOY study: UHN Umbrella Trial Defining Coordinated Approach to Pandemic Trials of COVID-19 and Data Harmonization to Accelerate Discovery. U-DEPLOY helps to facilitate timely conduct of studies across the University Health Network (UHN) and other centers.

DETAILED DESCRIPTION:
Given increasing community transmission and the possibility of asymptomatic carriage of virus, it is important to study whether asymptomatic shedders of virus are playing a role in propagating the pandemic. There is currently little data available regarding cancer patients, yet, this population may be particularly susceptible to the COVID-19 infection.

Despite the cancer patient population being at higher risk of COVID-19, no systematic screening has been established and no biomarkers have been identified to determine which patient is at higher risk.

This study will screen patients on active cancer therapy for COVID-19 as a standard of care or a research nasopharyngeal test. Blood samples may also be taken to assess any patient response to the virus and optional saliva samples may also be taken to assess the feasibility of using patient saliva for detection of SARS-CoV-2 virus in patients with impaired saliva production (eg. secondary to cancer treatments such as radiation, chemotherapy, and/or surgery).

ELIGIBILITY:
Inclusion Criteria:

* Patients having an active malignancy who are planned to start therapy within 6 weeks of consent or are receiving a treatment for active malignancy.
* The patient falls under either of the following categories:

  1. Asymptomatic for COVID-19 (as per daily screening at the hospital entrance).
  2. Has symptoms similar to those of COVID-19 (e.g. fever or flu-like symptoms such as cough or shortness of breath) that are assessed by the overseeing Investigator as being related to disease and unrelated to COVID-19 infection.

Note: Patients who recovered from previous COVID-19 infection will be eligible.

* No contraindication to performing a NP swab and blood work.

Exclusion Criteria:

* Any patients with fever, or flu-like symptoms assessed by the Investigator to be related or potentially related to COVID-19 infection will not be eligible.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 3-4

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients having an active malignancy who are planned to start therapy or receiving a treatment for active malignancy involved at the University Health Network and any other centres that choose to participate that are asymptomatic to COVID-19 for in-patients or ambulatory patients.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
Rate of asymptomatic COVID-19 infection among cancer patients receiving cancer therapy | 12 months

SECONDARY OUTCOMES:
Rate of sero-conversion in cancer patients | 12 months
Describe the clinical course of COVID-19 infection in cancer patients | 12 months

OTHER OUTCOMES:
Feasibility of using patient saliva for detection of SARS-CoV-2 virus in patients with impaired saliva production | 12 months
Compare the evolution of immune and proteomic profile of asymptomatic COVID-19 negative and positive cancer patients | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lheureux, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada